CLINICAL TRIAL: NCT03979456
Title: RItuximab Long-Term DOSE Trial in Multiple Sclerosis - RIDOSE-MS. A Randomized Trial of Long-term Dosage of Rituximab in Multiple Sclerosis
Brief Title: RItuximab Long-Term DOSE Trial in Multiple Sclerosis - RIDOSE-MS
Acronym: RIDOSE-MS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Svenningsson, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT 2018-000721-31
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple sclerosis; Relapsing-Remitting; Dosing protocols; Randomized trial
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Rituximab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 6-month dosing interval (Active Comparator): This arm is receiving standard dose rituximab 500 mg every 6 months
  Interventions: Drug: Rituximab
- 12-month dosing interval (Experimental): This arm is receiving the comparator dose rituximab 500 mg every 12 months
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — After one year in the trial, the patients are split in the two dosing-arms described above. The dose-comparison phase continues four years.
  Other Names: Mabthera

SUMMARY:
A randomized trial of long-term dosage of rituximab in multiple sclerosis

DETAILED DESCRIPTION:
This is a prospective randomized phase 3 study comparing two dosing regimens of Rituximab in long-term treatment of MS. Primary endpoint is no evidence of disease activity (NEDA) in a non-inferiority analysis between 12-months dosing interval of 500 mg rituximab with 6-months dosing interval. The endpoint is a compound of being free from release, new or enlarging MRI lesions and sustained progression of disability measured by EDSS.

Each patient will have one treating physician responsible for all ongoing medical questions and decisions regarding continuation in the study and one examining physician performing the blinded Expanded Disability Status Scale examination and assessments of exacerbations. The coordinating nurse will administer the study-related tests and administer the rituximab infusions. MRI investigations will be performed blinded for the dosing arm allocation.

Randomization will be performed via a randomization module in the national Swedish MS registry. The patients will be randomized in a 1:1 ratio and receive their treatments in accordance with clinical practice. Thus, the study will mimic the real-life situation in which the treatments will be administered. This will lead to a high degree of validity in relation to expected outcome in clinical practice.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of Relapsing Remitting MS according to the 2017 revised McDonald criteria OR one demyelinating episode in conjunction with at least one asymptomatic high intensity T2 lesion with size and location compatible with MS
* The patient has completed the RIFUND-MS trial and is treated with either of the study medications rituximab or DMF at the last visit of the RIFUND trial OR has been treated with rituximab with a dose regimen of 500 - 1000 mg followed by 500 mg every 6 months for up to two years as part of clinical practice
* Age 20 - 52 years (inclusive)
* EDSS 0 - 5,5 (inclusive)
* The patient is willing and able to give written informed consent, according to the judgement of the investigator.
* In fertile females, willing to comply with effective contraceptive methods. These include birth control pills, surgical sterilization of patient or partner or intrauterine device. Non-fertile women is defined as more than 12 months of amenorrhea without an alternative medical cause or, in case of ambiguities, an FSH level in the postmenopausal range.

Exclusion criteria:

* Diagnosis of Progressive MS
* Previous treatment with any "second-line" immunomodulatory drug, eg natalizumab, alemtuzumab, fingolimod, or other long-acting immunosuppressive agents.
* Pregnant or lactating women s-HCG will be tested on all women at screening, before each study-related infu-sion and in any situation where there is a reason to suspect pregnancy during the trial, e.g delayed menstrual period more than five days above expected time.
* Patients having contraindication for or otherwise not compliant with MRI investigations
* Simultaneous treatment with other immunosuppressive drugs
* Active, severe infections Signs of infections are assessed before inclusion and each study-related infusion through clinical examination and further evaluated by laboratory and other relevant investigations in case of suspected ongoing infection. Hepatitis serology (HBsAg and anti-HBc) will be evaluated before treatment onset if not tested within the previous three years.
* Severe cardiac disorder, e.g signs of congestive heart failure or coronary artery disease. This will be evaluated through clinical assessment before inclusion.
* Vaccination within 4 weeks of first dose of study medication.
* Documented allergy or intolerance to the IP
* Severe psychiatric condition

Ages: 20 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-04 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
No evidence of disease activity (NEDA) | 3 years
  The proportion of patients maintaining No Evidence of Disease Activity-3 (NEDA-3) during year 2 - 4 of the trial: No relapse, no new T2 lesions (> 3 mm), no EDSS progression in either dose arm

SECONDARY OUTCOMES:
No evidence of disease activity (NEDA) in subgroups | 4 years
  The proportion of patients maintaining NEDA-3 comparing the previous rituximab arm with the previous DMF arm from the RIFUND trial
Time to first relapse | 3 yeas
  Time to first relapse for the two dose arms
Freedom of new or enlarged lesions on MRI | 3 years
  Proportion of patients in each dosing arm without new/enlarging T2 lesions
Development of brain atrophy | 3 years
  Evolution of brain atrophy measured as brain parenchymal fraction (BPF) and corpus callosum area or -volume
Development of confirmed sustained disability | 3 years
  Proportion of patient with confirmed progression in EDSS according to pre-specified criteria
Mean progression of disability | 3 years
  The mean change in EDSS over the trial period in the two dosing arms
Neurodegeneration | 3 years
  The mean change of s-NFL concentration between the two dosing arms
Dose persistence | 3 years
  Time to discontinuation of dosing regimen allocation
Development of hypogammaglobulinaemia | 3 years
  The occurrence of hypogammaglobulinaemia in the two dosing arms
Development of neutropenia | 3 years
  The occurrence of neutropenia in the two dosing arms
Development of infections | 3 years
  The occurrence of infections in the two dosing arms

OTHER OUTCOMES:
Health economy | 3 years
  Estimation of societal costs per year to supply the two dosing arms
Treatment Satisfaction Questionnaire | 3 years
  Validated scale that evaluate the degree of treatment satisfaction through 10 5- or 7 grade likert-scale questions

CONTACTS AND LOCATIONS:
Overall Officials: Anders Svenningsson, Professor, Principal Investigator — Dept of Clinical Sciences, Karolinska Institutet Danderyd Hospital, Stockholm
Locations (17):
- Sweden (17):
  - Anders Svenningsson, Danderyd, Stockholm County
  - South Älvsborg Hospital, Borås
  - Falun Hospital, Falun
  - Gävle Hospital, Gävle
  - Saghlgrenska Hospital, Gothenburg
  - Helsingborg Hospital, Helsingborg
  - Karlstad Hospital, Karlstad
  - Halland Hospital Kungsbacka, Kungsbacka
  - Linköping University Hospital, Linköping
  - Nyköping Hospital, Nyköping
  - Örebro University Hospital, Örebro
  - Östersund Hospital, Östersund
  - Capio StGöran Hospital, Stockholm
  - Fredrik Piehl, Stockholm
  - Karolinska Hospital Huddinge, Stockholm
  - Umeå University, Umeå
  - Uppsala Academiska Hospital, Uppsala